CLINICAL TRIAL: NCT03784170
Title: Evaluation of a Non-Implanted Electrical Stimulation Continence Device for Overactive Bladder
Brief Title: FemPulse Therapy for Overactive Bladder in Women
Acronym: EVANESCE-OAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FemPulse Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIP-002
Record Dates: First submitted 2018-12-14; First posted 2018-12-21 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2020-02

CONDITIONS: Urinary Bladder, Overactive
Keywords: Overactive Bladder; OAB; Women; Neuromodulation; Bioelectronic Medicine
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: Subjects will wear a device and will be treated at 1 of 2 device settings for approximately 3 days.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Treatment (Experimental): FemPulse System at one device setting
  Interventions: Device: FemPulse System
- Control (Sham Comparator): FemPulse System at a different device setting
  Interventions: Device: FemPulse System

INTERVENTIONS:
Device: FemPulse System — Device therapy with the FemPulse System

SUMMARY:
The purpose of this clinical trial is to investigate a new medical device treatment for Overactive Bladder (OAB) in women.

DETAILED DESCRIPTION:
The FemPulse System is a vaginal ring intended to provide mild electrical stimulation to nerves that regulate bladder function. It is believed that stimulation of these nerves may help relieve the symptoms of OAB.

ELIGIBILITY:
Inclusion Criteria:

* Females 21 years or older with a diagnosis of Overactive Bladder
* If of reproductive age, must use a reliable form of contraception

Exclusion Criteria:

* Pregnant, was recently pregnant or is trying to conceive
* Has a metal pelvic implant or any electrically active implanted medical device
* Had a previous hysterectomy, pelvic radiation or pelvic cancer
* Has significant pelvic organ prolapse
* Had bladder treatment with onabotulinumtoxinA in the previous 12 months
* Has a significant heart condition

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
All device- and procedure-related adverse events will be collected and tabulated | Approximately 11 days in total
  Adverse events
Urinary frequency | Approximately 11 days in total
  Frequency of and intervals between urinary voids (voids per day and time between voids)
Urinary urgency | Approximately 11 days in total
  Presence or absence of urgency with each void
Urge urinary incontinence (UUI) | Approximately 11 days in total
  Presence or absence of UUI with each void
OAB-q - Short Form | Approximately 11 days in total
  OAB bother quality of life questionnaire
OAB Symptom Score | Approximately 11 days in total
  OAB symptoms quality of life questionnaire
Urogenital Distress Inventory - Short Form | Approximately 11 days in total
  OAB-related distress quality of life questionnaire
Incontinence Impact Questionnaire - Short Form | Approximately 11 days in total
  Impact of OAB quality of life questionnaire

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Minnesota Urology, Woodbury, Minnesota
  - McKay Urology, Charlotte, North Carolina
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No